CLINICAL TRIAL: NCT02535429
Title: Massage Therapy for HIV-positive People : Effects on Anxiety, Depression, Hyperventilation and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HIV massage
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: HIV-positive Diagnosis
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- massage (Experimental): massage
  Interventions: Other: massage
- Control (No Intervention)

INTERVENTIONS:
Other: massage
  Arms: massage

SUMMARY:
Massage therapy during 1 month and evaluation of depression, hyperventilation, anxiety and quality of life

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive diagnosis

Exclusion Criteria:

* musculoskeletal disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Anxiety measured by Hospital anxiety and depression scale | 5 minutes
Depression measured by Hospital anxiety and depression scale | 5 minutes
Hyperventilation measured by NIJMEGEN questionnaire | 5 minutes
quality of life measured by World Health Organization Quality of Life Questionnaire | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique universitaire Saint-Luc, Brussels, Belgium